CLINICAL TRIAL: NCT04433832
Title: Epidemiology and Prognostic Implications of Panic Disorder and Generalized Anxiety Disorder in Patients With Coronary Artery Disease
Brief Title: Physical and Psychological Health Trajectories in the Context of Coronary Heart Disease
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Laval University (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government); Quebec Heart Institute (Other); CISSS de Chaudière-Appalaches (Other Government)
Responsible Party: Principal Investigator, Guillaume Foldes-Busque, Professor, Laval University
Other Study IDs: LavalU
Record Dates: First submitted 2020-05-28; First posted 2020-06-16 (Actual); Last update posted 2020-10-30 (Actual); Status verified 2020-10

CONDITIONS: Panic Disorder; Generalized Anxiety Disorder; Coronary Artery Disease; Anxiety Disorders
Keywords: Coronary artery disease; Anxiety; Anxiety disorders; Prognosis; Cardiac rehabilitation; Psychosocial risk factors; Health behaviors; Treatment adherence
MeSH Terms: conditions — Panic Disorder; Generalized Anxiety Disorder; Coronary Artery Disease; Anxiety Disorders; Health Behavior; Treatment Adherence and Compliance

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The primary aim of this study is to establish how frequently patients with coronary artery disease present or develop two anxiety disorders (panic disorder and generalized anxiety disorder) in the two years following a medical intervention for their heart. A second objective is to assess the impact of these anxiety disorders on the health of these patients.

DETAILED DESCRIPTION:
Coronary artery disease (CAD), the most common form of cardiovascular disease, affects approximately 1 in 12 adults in Canada. CAD is a major public health concern and is one of the costliest chronic diseases in North America. Up to 90% of the CAD risk is attributable to nine modifiable risk factors, including psychosocial factors. Decades of research confirmed the importance of psychosocial factors in the development, prognosis and clinical presentation of CAD. One understudied but highly significant psychosocial risk factor is anxiety. Prevalence estimates of anxiety disorders in patients with CAD range from 10% to 65%, with panic disorder (PD) and generalized anxiety disorder (GAD) being the most prevalent. Both PD and GAD have been independently associated with a 36% to 94% increase in the risk of adverse cardiac events in patients with CAD. However, these findings remain controversial as some studies reported either an inverse or no association between PD and adverse events. Still, both PD and GAD are associated with the presence of multiple risk factors for CAD (e.g. smoking, high alcohol consumption and a sedentary lifestyle). These anxiety disorders are also likely to influence medication taking behaviors as well as adherence to cardiac rehabilitation programs. These data highlight the importance and prognostic significance of PD/GAD in patients with CAD. However, considering the contradictory data and significant methodological issues in the available studies, notably in terms of the validity of PD and GAD diagnoses, new, methodologically sound studies are needed to improve our understanding of this clinical problem and improve patient care.

The primary aim of this study is to establish the prevalence and incidence of PD and GAD in the two years following a revascularization procedure for CAD. The secondary aim is to prospectively assess the association between these disorders and cardiac mortality, adverse cardiac events, adherence to recommended treatments (exercise, cardiac rehabilitation, pharmacotherapy),quality of life and psychological distress.

This prospective cohort study will include 3610 patients who will be consecutively recruited following a revascularisation procedure for CAD at the cardiology department of the Quebec Heart and Lung Institute. Patients will be assessed at baseline (within a week of admission) as well as 3, 6, 12 and 24 months later. PD and GAD will be assessed with a standardized and validated semi-structured interview. The presence of adverse events, adherence to treatments, psychological distress and quality of life will be assessed through a review of medical records, questionnaires and interviews.

ELIGIBILITY:
Inclusion Criteria:

* All adult patients (18 years of age or older) who undergo a revascularization procedure for CAD at the Quebec Heart and Lung Institute and who write/speak French will be eligible for study participation.

Exclusion Criteria:

* Patients will be excluded if they present a severe communication problem or suffer from a terminal illness, a diagnosed major cognitive deficit, or any other condition that could invalidate the interview (e.g. psychotic disorder).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults patients who write and speak French and who have undergone a revascularization procedure (percutaneous coronary intervention or coronary bypass grafting) for CAD.
Sampling Method: Probability Sample
Enrollment: 3610 (Estimated)
Dates: Start 2020-01-20 (Actual); Primary Completion 2022-06-30 (Estimated); Study Completion 2023-11-30 (Estimated)

PRIMARY OUTCOMES:
Anxiety and Related Disorders Interview Schedule for DSM-5 | 2 years
  Panic disorder (PD) and generalized anxiety disorder (GAD) will be assessed at each time point using the Anxiety and Related Disorders Interview Schedule for DSM-5 (ADIS-5). This standardized interview protocol is one of the recommended measures for diagnosing anxiety disorders, including PD and GAD, in the research context. The PD and GAD modules of previous versions of the ADIS have demonstrated excellent reliability for their respective diagnoses.
Adverse cardiac events | 2 years
  Patients will be asked about all potential adverse events during a structured medical interview developed by our team. All data will be confirmed by a review of medical records. With written permission from patients or next of kin (if deceased), records for admissions or consultations outside of the study hospitals will be obtained from the establishment archives. Medical data will be extracted by the research nurses using a standardized medical data extraction form known for its excellent reliability.
  Adverse events are defined as: either an acute myocardial infarction, a revascularization procedure (percutaneous coronary intervention or coronary bypass grafting), a cardiac arrest (including ventricular fibrillation) or death from a cardiovascular cause (primary cause).

SECONDARY OUTCOMES:
Medical Outcomes Study Measures of Patient Adherence | 2 years
  A 5-item general measure which assesses the patients' tendency to comply with medical recommendations and a second section which measures adherence to recommendations made by a healthcare professional (e.g., taking medication, following a diet) in the context of CAD. Total scores range from 0 to 25, higher scores indicate higher reported medication adherence.
Adherence Scale in Chronic Diseases | 2 years
  This measure specifically assesses medication adherence and some of its potential barriers in patients with CAD or other chronic diseases. Total scores range from 0 to 32, higher scores indicate higher reported medication adherence.
Cardiac rehabilitation participation | 2 years
  Patients will be asked if they participated in a formal rehabilitation program at each time point with two validated interview items. Attendance will be assessed by reviewing records of the 12-week cardiac rehabilitation programs. With written permission from patients or next of kin, records of attendance to programs outside of the study hospitals will be obtained from archives departments. Participation will be categorized as follows:
  * Non-attendance: patients who did not attend a cardiac rehabilitation program.
  * Level of adherence: calculated with the percentage of the prescribed sessions attended during the program.
  * Completion: patients who attended at least 70% of the planned sessions.
  * Discontinuation: patients who stopped attending cardiac rehabilitation at least 3 weeks before the end of the program.
Health behaviors - Level of physical activity | 2 years
  Level of physical activity: This parameter will be assessed with the validated French version of the International Physical Activity Questionnaire - Short Form. This questionnaire generates an average amount of time spent per week doing physical activity across activity domains. A higher mean time represents more physical activity on average.
Health behaviors - Smoking status | 2 years
  Smoking status: This variable will be assessed using the validated self-report items developed by Statistics Canada to assess the current smoking status. Smoking status will be established based on the patients' self-reported smoking behaviour in the 30 days preceding each time point. Participants can be categorized as Non-Smokers, Occasional-Smokers or Regular Smokers.
Health behaviors - Alcohol use | 2 years
  Alcohol use: The patients' compliance with recommendations regarding alcohol consumption will be assessed with the first 3 items of the validated French version of the Alcohol Use Disorders Identification Test. Total scores range from 0 to 12, higher scores indicate higher alcohol use.
Health behaviors - Fruit and vegetable intake | 2 years
  Fruit and vegetable intake: Patients' usual consumption of fruit and vegetables will be assessed using the 6-item Fruit and Vegetable Questionnaire (FV-Q) validated questionnaire. This questionnaire generates a mean daily consumption of fruits and vegetables. A higher mean represents more servings consumed for each specific category.
Quality of life and psychological distress - Health-related quality of life | 2 years
  Health-related quality of life: The 12-item Short-Form Health Survey Version 2 (SF-12v2) will be used to assess patients Health-related quality of life.
  Total scores range between 0 and 100, with higher scores indicating a better HRQOL.
Quality of life and psychological distress - Anxiety and depressive symptoms | 2 years
  Anxiety and depressive symptoms will be measured with the validated French version of the Hospital Anxiety and Depression Scale.
  Total scores range between 0 and 21, with higher scores indicating a higher level of anxiety/depression.
Quality of life and psychological distress - Heart- focused anxiety | 2 years
  Heart- focused anxiety will be assessed with the French version of the Cardiac Anxiety Questionnaire. Total scores range between 0 and 20, with higher scores indicating a higher level of heart-focused anxiety.
PTSD Checklist for DSM-5 | 2 years
  The PCL-5 is a 20-item self-report questionnaire that assesses post-traumatic stress disorder (PTSD) symptoms according to DSM-5 criteria. In this study, the PCL will be used to assess symptom severity and to make a provisional PTSD diagnosis.
  Total scores range between 0 and 80, with higher scores indicating a higher level of PTSD.

OTHER OUTCOMES:
Sociodemographic data | 2 years
  Sociodemographic information, including employment status, educational level and family income (i.e. socio-economic status), will be obtained using a brief questionnaire.
Medical comorbidities and medical risk factors for CAD | 2 years
  These data will be obtained through a medical interview and structured review of medical records. Obesity will be assessed using body mass index, which will be computed from the reported height and weight of patients obtained during the medical interview (kg/m2).
Other psychosocial risk factors for CAD - Social support | 2 years
  Social support will be assessed with the validated French version of the Modified MOS Social Support Survey. This questionnaire generates two distinct subscales, emotional and instrumental support. Each subscale score ranges from 0 to 20, with higher scores representing more perceived support.
Other psychosocial risk factors for CAD - Depression, agoraphobia, health anxiety and somatic symptom disorders | 2 years
  Depression, agoraphobia, health anxiety and somatic symptom disorders will be assessed with the ADIS-5.

CONTACTS AND LOCATIONS:
Overall Officials: Guillaume Foldes-Busque, Ph.D., Principal Investigator — Laval University
Locations (1):
- Quebec Heart and Lung Institute/Institut universitaire de cardiologie et de pneumologie de Québec, Québec, Canada

IPD SHARING:
Plan to Share IPD: No